CLINICAL TRIAL: NCT05974982
Title: Comparison of the Outcome of Treatment With Autologous Platelet Rich Plasma Versus Conventional Therapy for Patients Presenting With Chronic Venous Leg Ulcers
Brief Title: Treatment Outcome of Autologous PRP Versus Conventional Therapy Among Patients With Chronic Venous Leg Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Faiza Inam Siddiqui, Resident dermatologist (fcps), Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.F.2-81/2022-GENL/249/JPMC
Record Dates: First submitted 2023-07-11; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich plasma (Experimental): Under aseptic precautions 20 ml of venous blood was drawn and added to a test tube containing acid citrate dextrose in a ratio of 9:1 (blood: Acid citrate dextrose), centrifuged at 5000 rpm for 15 min to separate the red blood cells from the platelets and plasma. Then the supernatant and the buffy coat composed of platelets and plasma were collected and centrifuged again at 2000 rpm for 5-10 min. The bottom layer about 1.5 ml was taken and 10% calcium chloride was added (0.3 ml for 1 ml of PRP). Then the activated PRP was applied to the wound after proper surgical debridement and was dressed with a non-absorbent dressing (paraffin gauze). This process was repeated once weekly for 6 weeks.
  Interventions: Biological: PRP
- Conventional therapy (Active Comparator): These patients were treated conservatively by compression using graduated elastic stockings below the knee and dressing using saline and vaseline gauze weekly for 6 weeks.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Biological: PRP — PRP is a volume of autologous plasma that has a platelet concentration above baseline i.e., five times more than normal platelet counts. PRP enhances wound healing by promoting the healing process by seven growth factors present in it. They are platelet derived growth factor (αα, αβ, αβ), fibroblast growth factor, vascular endothelial growth factor, epidermal growth factor, transforming growth factor.
  Arms: Platelet-rich plasma
Other: Conventional therapy — Conventional therapy
  Arms: Conventional therapy

SUMMARY:
The use of PRP has dramatically increased in the fields of orthopedics, spine surgery, reconstructive plastic surgery, oral and maxillofacial surgery, and dermatological indications. Nonetheless, its use in the treatment of wounds is not as widespread as in other fields. In this experimental study, the treatment outcome of autologous PRP was assessed in comparison to conventional therapy among patients with chronic venous leg ulcers.

DETAILED DESCRIPTION:
Venous ulcers are the most common form of leg ulcers which have a significant impact on quality of life and work productivity. In addition, the costs associated with the long-term care of these chronic wounds are substantial. Conventional therapies such as dressings, surgical debridement, compression bandage, and even skin grafting cannot provide satisfactory healing since these treatments are not able to provide necessary growth factors that can modulate healing processes. Autologous platelet-rich plasma (PRP) is a safe, simple, affordable, and less expensive procedure in the treatment of chronic ulcers with reportedly good results. Since it is an autologous method, it is biocompatible and safe. Data from this would help in establishing it as a treatment of choice, thereby leading to a reduction in cost and benefiting the patient both financially and psychologically.

PRP is a volume of autologous plasma that has a platelet concentration above baseline i.e., five times more than normal platelet counts. PRP enhances wound healing by promoting the healing process by seven growth factors present in it. They are platelet-derived growth factor (αα, αβ, αβ), fibroblast growth factor, vascular endothelial growth factor, epidermal growth factor, and transforming growth factor. These growth factors are important in modulating mesenchymal cell recruitment, proliferation, and extra-cellular matrix synthesis during the healing process.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-80 years of any gender presented with chronic venous leg ulcers

Exclusion Criteria:

* Patients with history of peripheral arterial disease.
* Patients with history of acute venous thromboembolism.
* Patients with platelet count less than 150000.
* Patients with history of bleeding disorders.
* Patients with history of osteoporosis.
* Patients with history of peripheral neuropathy.
* Pregnant patients assessed by history and confirmed by dating scan.
* Patients with history of congestive cardiac failure, chronic liver disease, asthma, COPD, or stroke.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Complete healing | 9 months
  Complete healing is defined as 100% epithelialization
Length of ulcer | 9 months
  Length of ulcer in cm at the end of treatment
Width of ulcer | 9 months
  Width of ulcer in cm at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ghafoor, Study Director — Jinnah Post Graduate Medical Centre
Locations (1):
- Jinnah Post graduate Medical centre, Karachi, Sindh, Pakistan